CLINICAL TRIAL: NCT05018429
Title: Nerve Sparing Versus Non Nerve Sparing Robot-assisted Radical Cystectomy-orthotopic Ileal Neobladder for Bladder Cancer in the Male
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Shantou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SysMU-RARC5
Record Dates: First submitted 2021-07-09; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nerve sparing group: Patients will be preverved the neurovascular bundles during the resection of bladder and prostate of the operation.
  Interventions: Procedure: nerve sparing
- non nerve sparing group: Patients will receive standard radical cystectomy (not preserve the neurovascular bundles) during the operation.

INTERVENTIONS:
Procedure: nerve sparing — When resect the bladder and prostate, the neurovascular bundles around the prostate will be preserved.
  Groups: nerve sparing group

SUMMARY:
To compare the perioperative, functional, and oncologic outcomes between non nerve sparing and nerve sparing robot-assisted radical cystectomy with orthotopic ileal neobladder in male patients with bladder cancer.

DETAILED DESCRIPTION:
This study will enroll male patients with bladder cancer who will undergo robot-assisted radical cystectomy with orthotopic ileal neobladder. The patients will be distributed into two comparable groups according to surgical procedures: non nerve sparing group and nerve sparing group. Patient demographic and pathologic, perioperative, functional, and oncologic outcomes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged 18 or older.
2. Patients those who are diagnosed with urothelial carcinoma.
3. Patients those who are capable of receiving radical cystectomy with orthotopic ileal neobladder.
4. Patients those who are able to cooperate and complete the follow-up.
5. Patients those who volunteer to participate in this study and sign the informed consens.

Exclusion Criteria:

1. Patients thsoe who are diagnosed distant metastasis before surgery.
2. Patients those who are diagnosed with other malignancies.
3. Patients those who had received pelvic radiotherapy or major pelvic operation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enroll patients who received RARC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
day-time continence rate | 6 months
  Patients were considered continent when they required 0 or 1 safety pad during the day-time.
night-time continence rate | 6 months
  Patients were considered continent when they required 0 or 1 safety pad during the night.
postoperative sexual function | 6 months
  The sexual function are evaluated by the International Index of Erectile Function-5 (IIEF-5).

SECONDARY OUTCOMES:
perioperative complication rate | 3 months
operative time | 24 hours
estimated blood loss | 24 hours
overall survival | 1 year
recurrence-free survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No